CLINICAL TRIAL: NCT02809144
Title: A Novel Combination of Peripheral Nerve Blocks for Patients Scheduled for Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Lars Marius Ytrebo, Professor, University Hospital of North Norway
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0472
Record Dates: First submitted 2015-05-25; First posted 2016-06-22 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Nerve Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nerve block (Other): One novel nerve block combination
  Interventions: Procedure: Nerve block

INTERVENTIONS:
Procedure: Nerve block — Nerve block: 31 ml ropivacaine 7.5 mg/ml (Lateral sagittal infraclavicular brachial plexus block) + 4 ml ropivacaine 5 mg/ml (suprascapular nerve block) + 5 ml ropivacaine 5 mg/ml (superficial cervical plexus block)

SUMMARY:
Interscalene block has been the traditional regional anesthesia for shoulder surgery and postoperative pain. However, the risk of phrenic nerve palsy and irreversible nerve injury have encouraged search for alternative methods.

DETAILED DESCRIPTION:
Analyzing block effects of the lateral sagittal infraclavicular brachial plexus block(posterior and lateral chord), the investigators found it affecting all shoulder relevant nerves , except for the suprascapular and the supraclavicular nerves.

Accordingly, by combining a superficial cervical plexus block, suprascapular nerve block and block of the posterior and lateral chords infraclavicularly, the investigators believe this novel combination would provide anesthesia for patients scheduled for shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for shoulder surgery.
* American Society of Anesthesiologist grad I-III,
* 18-70 years,
* BMI 20-35,

Exclusion Criteria:

* Pregnancy,
* coagulopathy,
* allergy to local anesthetics,
* atrioventricular block,
* peripheral neuropathy or drug-treated diabetes.
* Patients using anticoagulation other than acetylsalicylic acid or dipyridamol will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The need for general anaesthesia | Intraoperatively
  Investigators will record the number of patients who need to be converted to general anaesthesia

SECONDARY OUTCOMES:
Surgeons satisfaction with the working conditions | Intraoperatively
  Graded in a) Good and b) Poor

CONTACTS AND LOCATIONS:
Overall Officials: Lars Marius Ytrebø, MD PhD, Principal Investigator — University Hospital of North Norway
Locations (1):
- University Hospital of North Norway, Tromsø, Troms, Norway

IPD SHARING:
Plan to Share IPD: No